CLINICAL TRIAL: NCT05282524
Title: HATCH (Helping Adults Perform Transvaginal Exams Via Coaching at Home) Study: Protocol for Training Ultrasound Technologists to Conduct At-home, Remote Transvaginal Ultrasounds
Brief Title: Helping Adults Perform Transvaginal Exams Via Coaching at Home
Acronym: HATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turtle Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 011
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Women's Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Simulated patient (Experimental): Women recruited from a general population subject to inclusion/exclusion criteria, who will participate at a minimum four times in the study
  Interventions: Device: Transvaginal ultrasound performed by a woman herself (with remote healthcare professional supervision)
- Naive patient (Experimental): Women recruited from a general population subject to inclusion/exclusion criteria, who will participate only once in the study
  Interventions: Device: Transvaginal ultrasound performed by a woman herself (with remote healthcare professional supervision)

INTERVENTIONS:
Device: Transvaginal ultrasound performed by a woman herself (with remote healthcare professional supervision) — Imaging performed by woman on herself with remote healthcare professional (HCP) supervision. The ultrasound device used is cleared for HCP-supervised use in environments where healthcare is provided by trained HCPs. No changes to the design or manufacture have been made for this study.

SUMMARY:
To train ultrasound technologists (equivalently called sonographers) in remote ultrasound guidance.

To capture imaging of the gynecologic organs visible on home ultrasound and pertinent to clinical care, specifically the ovaries and uterus.

To train the independent readers, both obstetricians & gynecologists (OB/GYNs) and reproductive endocrinologists (REIs), who will evaluate home ultrasound images over time in subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over who have not gone through menopause (defined as no menstruation for at least 12 months, not explained by other causes)
* Women with body mass index (BMI) up to 40
* Women who speak English, assessed through screening questions
* Women with at least a high school degree or equivalent (e.g., General Educational Development (GED) or similar)
* Women located in Massachusetts
* Women who are able to safely receive delivery of the ultrasound scanner
* Women between cycle days 3 and 10 at the time of testing as a mitigation against potential inadvertent early fetal exposure; or intrauterine device (IUD) users who do not have a menses
* Women who have all three primary gynecological organs: left ovary, right ovary, and uterus

Exclusion Criteria:

* Women with BMI over 40
* Women who do not speak English natively or fluently
* Women who have recently given birth, and have had fewer than 3 postpartum menstrual cycles
* Women who have recently had a stillbirth or abortion more than 20 weeks (subject to the 3 postpartum menstrual cycles above). Miscarriages or abortions less than 20 weeks are subject to two wait cycles
* Women who are currently pregnant or may be pregnant
* Women who have had a hysterectomy or oophorectomy
* Women who have changed birth control within the current menstrual cycle. (One 'washout' cycle is required)
* Women with cancer of any pelvic organ
* Women who are not able to schedule an exam while meeting the requirements above prior to the end of the trial. For example, women who change birth control within the last cycle of the trial (and would require a 'washout cycle' that would delay trial close) or who are unable to schedule within the last few weeks of the trial after reasonable scheduling efforts have been made may be excluded.
* Women with disabilities are excluded only if their disability precludes their ability to manipulate an ultrasound and follow technologist instructions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Video quality of remote self-performed ultrasound exam | 1 visit (up to 1 hour)
  Determination of whether each organ view is 'diagnostic quality' or 'not diagnostic quality' based on American Institute of Ultrasound in Medicine (AIUM) criteria/guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual metasite, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No